CLINICAL TRIAL: NCT04981015
Title: Bladder Diary Can be a Good Surrogate of Diagnosing Bladder Oversensitivity
Brief Title: Bladder Diary for Diagnosing Bladder Oversensitivity
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202105069RINA
Record Dates: First submitted 2021-07-20; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Bladder Oversensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with lower urinary tract symptoms: Women with lower urinary tract symptoms without cystocele were included.
  Interventions: Diagnostic Test: Three-day bladder diary

INTERVENTIONS:
Diagnostic Test: Three-day bladder diary — A three-day bladder diary for recording voiding-flow pattern of a women
  Other Names: Urodynamic study

SUMMARY:
Urodynamic study is an invasive procedure and applied for diagnosis of bladder oversensitivity. Bladder diary is a non-invasive measurement. The aim of this study was to elucidate whether bladder diary is a good surrogate for diagnosing bladder oversensitivity.

DETAILED DESCRIPTION:
Between July 2009 and December 2020, medical records of all women with lower urinary tract symptoms but without cystocele who visited the urogynecological department of a medical center for urodynamic evaluation were reviewed. Those women who have no complete data of a 3-day bladder diary were excluded from this study. Bladder oversensitivity was diagnosed if the volume of strong desire was less than 300mL. We compared the urodynamic parameters to bladder diary parameters in order to find the best correlation between these 2 measurements for the diagnosis of bladder oversensitivity.

STATA software was used for statistical analysis. Chi2 test, univariate and multivariable logistic regression tests were used for statistical analysis as appropriate. A p < 0.05 was considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Women with lower urinary tract symptoms
* Complete a urodynamic study
* Complete a 3-day bladder diary

Exclusion Criteria:

* Women with cystocele
* Chronic infection
* Incomplete data

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women with lower urinary tract symptoms but without cystocele who visited the urogynecological department of a medical center for urodynamic evaluation were included.
Sampling Method: Non-Probability Sample
Enrollment: 3960 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation between parameters | July 2009 to December 2020
  Correlation between 3-day bladder diary and urodynamic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Hsiung Lin, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data is available under reasonable request

REFERENCES:
- [Result] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Result] Coyne KS, Wein AJ, Tubaro A, Sexton CC, Thompson CL, Kopp ZS, Aiyer LP. The burden of lower urinary tract symptoms: evaluating the effect of LUTS on health-related quality of life, anxiety and depression: EpiLUTS. BJU Int. 2009 Apr;103 Suppl 3:4-11. doi: 10.1111/j.1464-410X.2009.08371.x. PMID 19302497
- [Result] Hsiao SM, Lin HH. Medical treatment of female overactive bladder syndrome and treatment-related effects. J Formos Med Assoc. 2018 Oct;117(10):871-878. doi: 10.1016/j.jfma.2018.01.011. Epub 2018 Feb 15. PMID 29398096
- [Result] Hsiao SM, Su TC, Chen CH, Chang TC, Lin HH. Autonomic dysfunction and arterial stiffness in female overactive bladder patients and antimuscarinics related effects. Maturitas. 2014 Sep;79(1):65-9. doi: 10.1016/j.maturitas.2014.06.001. Epub 2014 Jun 20. PMID 25022469
- [Result] Hsiao SM, Liao SC, Chen CH, Chang TC, Lin HH. Psychometric assessment of female overactive bladder syndrome and antimuscarinics-related effects. Maturitas. 2014 Dec;79(4):428-34. doi: 10.1016/j.maturitas.2014.08.009. Epub 2014 Sep 3. PMID 25238744